CLINICAL TRIAL: NCT03039322
Title: Golgi Protein 73 for Diagnosis of HCC in Egyptian Patients
Brief Title: Golgi Protein for HCC Diagnosis
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shereen Abou Bakr Saleh, Assisstant Professor, Ain Shams University
Other Study IDs: 914
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Screening for Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC
  Interventions: Diagnostic Test: Serum Golgi Protein 73
- liver cirrhosis No HCC
  Interventions: Diagnostic Test: Serum Golgi Protein 73

INTERVENTIONS:
Diagnostic Test: Serum Golgi Protein 73 — Serum test

SUMMARY:
This case-control study was conducted on 90 patients who were equally divided into two groups. Group 1 included 45 patients with HCV-related chronic liver disease without clinical or radiological evidence of HCC (control group), and Group 2 included 45 patients diagnosed to have HCC by Triphasic abdominal CT (patient group). Serum AFP and GP73 were measured using ELISA technique

ELIGIBILITY:
Inclusion Criteria:

* patients were older than 18 years.

Exclusion Criteria:

* patients with hepatic focal lesions not due to HCC such as Hemangioma, Hepatic cyst, and liver metastases; patients infected with HIV; patients with any autoimmune disease; or patients with metastatic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group I: Included 45 patients with liver cirrhosis due to HCV infection. Liver cirrhosis was diagnosed clinically, laboratory, and radiologically. Chronic HCV infection was diagnosed by positive HCV antibody and positive quantitative HCV PCR.
  Group II: Included 45 patients with Hepatocellular carcinoma (HCC) on top of HCV cirrhosis diagnosed by two imaging modalities, abdominal ultrasound and the characteristic arterial enhancement and venous washout in Tri-phasic CT abdomen.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Golgi protein correlated with presence of HCC | within one year